CLINICAL TRIAL: NCT03363516
Title: Early Prediction of Mild Cognitive Impairment in Glucose Normotolerant Subjects With 1-hour Post-load Plasma Glucose >155 mg/dL
Brief Title: 1-hour Post-load Hyperglycemia and Mild Cognitive Impairment
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Maria Perticone (Other)
Responsible Party: Sponsor-Investigator, Maria Perticone, Principal Investigator, University Magna Graecia
Organization: University Magna Graecia (Other)
Other Study IDs: UNICZ01
Record Dates: First submitted 2017-11-22; First posted 2017-12-06 (Actual); Last update posted 2017-12-07 (Actual); Status verified 2017-12

CONDITIONS: Glucose Metabolism Disorders; Mild Cognitive Impairment
MeSH Terms: conditions — Glucose Metabolism Disorders; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases: Glucose normotolerant subjects with 1-h post-load plasma glucose >155 mg/dL
  Interventions: Diagnostic Test: Cerebral 3 Tesla MRI
- Controls: Glucose normotolerant subjects with 1-h post-load plasma glucose <155 mg/dL
  Interventions: Diagnostic Test: Cerebral 3 Tesla MRI

INTERVENTIONS:
Diagnostic Test: Cerebral 3 Tesla MRI — Subjects will be examined using a 3 Tesla MR750 GE MRI scanner with an eight-channel head coil. All participants will undergo the same MRI protocol, including: whole-brain 3D T1-weighted spoiled gradient recalled (SPGR) (BRAVO, voxel size of 1 × 1 × 1 mm3), DTI (voxel size 2 × 2 × 2 mm3, 27 directions with gradients at a b-value of 1,000 s/mm2 and 4 b = 0 images) and conventional 2D T2-weighted,T2 (FLAIR) and T2 gradient echo.
  Other Names: Neuropsychological evaluation

SUMMARY:
Insulin resistance (IR), beyond its well-defined role in the appearance and progression of diabetes mellitus (DM), is the recognized pathogenetic factor underlying vascular aging. Recently, the existence of a "cerebral" IR, responsible of the appearance and progression of many forms of dementia and mild cognitive impairment (MCI), has been hypothesized. On the other hand, it is well known that DM acts as a cardiovascular (CV) risk factor per se. In the last years it has been demonstrated that also glucose normotolerant subjects who exhibit plasma glucose levels >155 mg/dL 1h-post load, have a CV risk similar to that of diabetic patients. Thus, these category of subjects is characterized by IR and, being MCI the expression of IR in the brain, the principal hypothesis of our study is that these subjects may also develop neuropsychological alterations, earlier with respect of the general population.

DETAILED DESCRIPTION:
Insulin resistance (IR), beyond its well-defined role in the appearance and progression of diabetes mellitus (DM), is the recognized pathogenetic factor underlying vascular aging, in the continuum from endothelial dysfunction to atherosclerotic vascular lesions. Two different types of IR have been described: 1) a "central" IR, particularly expressed in the liver, affecting all the metabolic pathways operating at this site, and 2) a "peripheral" IR, particularly expressed in the muscle. Recently, the existence of a "cerebral" IR, responsible of the appearance and progression of many forms of dementia and mild cognitive impairment (MCI), has been hypothesized. On the other hand, for decades DM was considered only as a hyperglycemic status, disregarding its important negative impact on vascular function and its role as a cardiovascular (CV) risk factor per se. For these reasons, in the past, DM management only consisted in reducing plasma glucose levels. In the last years our group demonstrated that also glucose normotolerant subjects who exhibit plasma glucose levels >155 mg/dL 1h-post load, have a CV risk similar to that of diabetic patients.

Hypothesis and Significance The hypothesis of this study is based on the concept that glucose normotolerant subjects with 1h-post load glycemia >155 mg/dL exhibit an insulin-resistant status characterized by enhanced insulin production but reduced tissues sensitivity to the hormone action. This reduced insulin sensitivity is present many years before the appearance of the clinical conditions such as DM, arterial hypertension, dyslipidemia, etc. Insulin, insulin receptor, and its substrates are expressed in the whole central nervous system; in this site, insulin regulates food intake and body weight, and it is also involved in neurotransmitters release and synaptic plasticity. It is thus plausible that insulin may have an important role in many cognitive processes. Evidences indicate that the cognitive impairment commonly seen in many diabetic patients could be mediated by an altered signaling insulin-like growth factor-1 (IGF1)-insulin. In fact, a stream of human and experimental studies has provided convincing evidence that many forms of dementia, such as Alzheimer's disease, are metabolic diseases characterized by the brain loss of its capacity to efficiently utilize glucose for energy production and respond to critical trophic factor signals due to insulin as well as insulin-like growth factor (IGF) resistance. Thus, being MCI the expression of IR in the brain, the principal hypothesis of our study is that these subjects may also develop neuropsychological alterations, earlier with respect of the general population. This hypothesis may have an important clinical significance and a great social impact, since a great amount of health costs are due chronic diseases, included all forms of dementia. Furthermore, the results of this study will add important information about the understanding of the complex network of pathways operating in the appearance and progression of many of the chronic diseases, such as diabetes mellitus and dementia.

Aim of the study To investigate the presence of early neuropsychological and/or cerebral morphological alterations in two groups of subjects (Group 1: glucose normotolerant subjects with 1h-post load glycemia >155 mg/dL; Group 2: healthy subjects with 1h post-load glycemia < 155 mg/dL).

Experimental Design

Visit 1: evaluation of inclusion/exclusion criteria, MMSE, clinical visit, all laboratory determinations, OGTT

Visit 2: neuropsychological assessment (refers to the measurement of cognitive functions and processes with the aim to establish whether a cognitive impairment is present in individuals. It is preferably performed by clinical neuropsychologists who have expertise in the study of the neural correlates of behavior and cognition. The cognitive processes to be investigated in the present study include functions such as memory, language, praxia, attention, executive functions and intelligence. The following tests will be used: MMSE, RAVLT, FCSRT, COWAT, FAB, TMT and Stroop Test, Weigl Test, BDI II, HAMA

3Tesla (T) brain magnetic resonance imaging (MRI) Subjects will be examined using a 3 Tesla MR750 GE MRI scanner with an eight-channel head coil. All participants will undergo the same MRI protocol, including: whole-brain 3D T1-weighted spoiled gradient recalled (SPGR) (BRAVO, voxel size of 1 × 1 × 1 mm3), DTI (voxel size 2 × 2 × 2 mm3, 27 directions with gradients at a b-value of 1,000 s/mm2 and 4 b = 0 images) and conventional 2D T2-weighted,T2 (FLAIR) and T2 gradient echo.

Methodologies and statistical analyses The investigators planned to conduct an observational perspective longitudinal study. The planned number of patients is 15 for each group. In particular, will be enrolled 15 glucose normotolerant subjects with 1h post-load glycemia >155 mg/dL (Group 1), and 15 healthy subjects with 1h post-load glycemia <155 mg/dL (Group 2).

All subjects will undergo the following study procedures:

* Clinical visit
* Measurement of vital signs
* Routine blood tests
* Oral glucose tolerance test (OGTT)
* Insulinemic curve
* Neuropsychological tests administration
* 3T brain MRI

Data will be collected in a case report form (CRF) mantained at the University Magna Graecia of Catanzaro. Data collected will be analyzed through descriptive statistic methodologies, t-test, ANOVA, linear and multiple regression, when appropriate.

Expected outcomes On the basis of previously published literature and of pathophysiologic hypothesis, the expected outcomes of this project are the early recognition of neuropsychological and/or neuroimaging alterations suggestive of mild cognitive impairment in insulin-resistant subjects without clinical evidence of metabolic diseases typical of the insulin-resistant status (diabetes mellitus, arterial hypertension, metabolic syndrome, etc.).

Significance and Innovation The results of this study could represent an important milestone in the comprehension of the complex pathophysiological mechanisms underlying the appearance of cognitive disorders in subjects with apparently different risk factors. If this hypothesis -that IR is the trait d'union between metabolic and cerebral alterations- will be confirmed, a new important link (i.e.: the relationship between IR/glucose metabolism and cerebral functions) could be further explored in future studies in order to plan preventive/therapeutic strategies for subjects with any type of insulin resistance, before the appearance of the clinical manifestations of IR in any of the target organs. The major innovation of this study is represented by the fact that IR could be considered not only as a cardiometabolic risk factor, but also as a cerebral one.

Translational relevance This study has an important scientific relevance since it is, to the investigators' knowledge, the first one merging both neuropsychological and metabolic aspects in a pre-clinical status. Thus, if the hypothesis of the study will be confirmed, the management of patients with IR could also include neuropsychological and neuroimaging assessments in order to early detect cognitive impairment.

ELIGIBILITY:
Inclusion Criteria:

* Subjects of both sex aged 55 years or older
* Ability to give informed written consent
* Mini mental state evaluation (MMSE) >20 at visit 1

Exclusion Criteria:

* Diabetes mellitus
* Clinically evident dementia or cognitive impairment
* Previous diagnosis of any disease predisposing to the risk of cognitive impairment (eg.: arterial hypertension, lipid metabolism alterations, obesity)
* Liver cirrhosis
* Family history of dementia and/or cognitive impairment
* History of alcohol or drugs abuse
* Use of medications influencing glucose homeostasis or cognitive functions
* Contraindications to undergo cerebral 3T-MRI
* Previous transient ischemic attack or stroke
* History of malignancies

Min Age: 55 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Subjects of both sexes, aged >55 yrs, afferent to our Internal Medicine Ward for cardio-metabolic risk factors screening
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2016-10 (Actual); Primary Completion 2018-09 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Evidence of early neuropsychological and/or cerebral morphological/functional alterations of MCI in cases | 1 month after enrollment
  Neuropsychological tests will be administered to all the study participants. All subjects will undergo an accurate evaluation of all the major cerebral functions in order to detect early alterations suggestive of mild cognitive impairment. Furthermore, all subjects will undergo a cerebral magnetic resonance using a 3 Tesla MR750 GE MRI scanner with an eight-channel head coil. All participants will undergo the same MRI protocol, including: whole-brain 3D T1-weighted spoiled gradient recalled (SPGR) (BRAVO, voxel size of 1 × 1 × 1 mm3), DTI (voxel size 2 × 2 × 2 mm3, 27 directions with gradients at a b-value of 1,000 s/mm2 and 4 b = 0 images) and conventional 2D T2-weighted,T2 (FLAIR) and T2 gradient echo. This test will investigate possible morphological and functional alterations suggestive of early dementia/MCI.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Perticone, Dr, Principal Investigator — University Magna Graecia of Catanzaro
Locations (1):
- University Magna Graecia of Catanzaro - Department of Medical and Surgical Sciences - Internal Medicine and Geriatrics Units, Catanzaro, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Willette AA, Bendlin BB, Starks EJ, Birdsill AC, Johnson SC, Christian BT, Okonkwo OC, La Rue A, Hermann BP, Koscik RL, Jonaitis EM, Sager MA, Asthana S. Association of Insulin Resistance With Cerebral Glucose Uptake in Late Middle-Aged Adults at Risk for Alzheimer Disease. JAMA Neurol. 2015 Sep;72(9):1013-20. doi: 10.1001/jamaneurol.2015.0613. PMID 26214150
- [Background] Willette AA, Xu G, Johnson SC, Birdsill AC, Jonaitis EM, Sager MA, Hermann BP, La Rue A, Asthana S, Bendlin BB. Insulin resistance, brain atrophy, and cognitive performance in late middle-aged adults. Diabetes Care. 2013 Feb;36(2):443-9. doi: 10.2337/dc12-0922. Epub 2012 Oct 15. PMID 23069842
- [Background] Kim B, Feldman EL. Insulin resistance as a key link for the increased risk of cognitive impairment in the metabolic syndrome. Exp Mol Med. 2015 Mar 13;47(3):e149. doi: 10.1038/emm.2015.3. PMID 25766618
- [Background] de la Monte SM. Type 3 diabetes is sporadic Alzheimer׳s disease: mini-review. Eur Neuropsychopharmacol. 2014 Dec;24(12):1954-60. doi: 10.1016/j.euroneuro.2014.06.008. Epub 2014 Jun 28. PMID 25088942